CLINICAL TRIAL: NCT04590053
Title: A Multi-Center Open-Label Study, Evaluating Safety and Preliminary Efficacy of Allocetra-OTS for the Treatment and Prevention of Organ-Failure Deterioration in Severe and Critical Patients With COVID-19 and Respiratory Dysfunction
Brief Title: Allocetra-OTS in COVID-19, Phase II
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Barzilai Medical Center (Other); Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Mevorach Dror, Professor & Head, Department of Internal Medicine B; Head, Rheumatology Research Center, Hadassah and the Hebrew University Medical School, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DM004
Record Dates: First submitted 2020-10-15; First posted 2020-10-19 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COVID-19 (Experimental): Up to 24 subjects, male or female > 18 and < 80-year-old diagnosed with respiratory dysfunction and COVID-19, as defined in the Eligibility Criteria, and treated with a single intravenous dose of Allocetra-OTS investigational product as detailed in the Interventions section.
  Interventions: Biological: Allocetra-OTS

INTERVENTIONS:
Biological: Allocetra-OTS — Allocetra-OTS is a cell-based therapeutic composed of donor early apoptotic cells, comprising allogeneic mononuclear enriched cell suspension with at least 40% early apoptotic cells. The suspension is prepared with Ringer's lactate solution and administered IV. It is stored at 2-8°C until 20+25 minutes before infusion and at room temperature thereafter. Each dose contains 140x10E6 ± 20% cells/ kg of recipient body weight (at screening) in a total volume of 375 mL in a transfer pack that undergoes irradiation and is administered via an adjusted filter using a volumetric pump, at a starting rate of 48 mL/hour with a gradual increase every 15-25 minutes of 15 mL/hour to a maximal rate of 102 mL/hour. The study intervention should be completed within 72 hours of completing the manufacturing process. During product administration, no other IV fluids such as Ringer's lactate or normal saline will be given in parallel unless medically indicated due to volume depletion.

SUMMARY:
This is a multi-center, open-label study evaluating the safety of Allocetra-OTS, in up to 24 subjects with severe COVID-19 and respiratory dysfunction. Subjects, who will be identified as suffering from COVID-19, will be recruited.

After signing an informed consent by the patient and, within 24+6 hours following the time of eligibility (time 0), on Day 1, eligible recipient subjects will receive single intravenous (IV) administration of investigational product as described below.

Subjects will be hospitalized for COVID-19, and later as medically indicated. Following the investigational product (IP) administration (Day 1), subjects will be followed for efficacy and safety assessments through 28 days.

DETAILED DESCRIPTION:
Study Rationale

COVID-19, the name given to the clinical syndrome associated with the newly recognized virus SARS-CoV-2, has become pandemic with a mortality estimated between 1-4% and complications among hospitalized patients leading to up to 15-25% of hospital admissions being admitted to the intensive care unit (ICU).

The term "cytokine storm" calls up vivid images of an immune system gone awry and an inflammatory response flaring out of control. The term has captured the attention of the public and the scientific community alike and is increasingly being used in both the popular media and the scientific literature. Indeed, a few publications have indicated an important part of the complications in COVID-19 are related to the cytokine storm (Huang et al. Lancet 2020, Mehta et al. Lancet 2020).

In a clinical study conducted in sepsis patients with Allocetra-OTS (ClinicalTrials.gov Identifier: NCT03925857) we observed that administration of Allocetra-OTS to patients with sepsis was safe and had a significant immuno-modulating effect, leading to resolution of the cytokine storm in these patients. There were indications that this treatment may also be efficacious, based on comparisons with mortality score prediction and historical matched-controls, and the resolution of organ dysfunction compared to matched historical controls.

A recent study published by Zou et al (Lancet 2020) showed increasing odds of in-hospital death in these COVID-19 patients associated with older age and higher Sequential Organ Failure Assessment (SOFA) score on admission.

Taken together, in patients with severe COVID-19, there may be a comparable underlying immunological mechanism of action as was recently demonstrated by us in sepsis; that is a hyper-inflammatory pathway associated with increased death. Therefore, a study of 5 patients was designed to determine the safety of this treatment in patients with severe COVID-19 and was approved by the Ministry of Health Ethical Committee. Based on the approved protocol, the intermediate clinical results of this trial show that the drug is safe and promising.

Study Design

This is a multi-center, open-label study evaluating the safety of Allocetra-OTS, in up to 24 adult patients with severe COVID-19 and respiratory dysfunction. Subjects, who will be identified as suffering from COVID-19, will be recruited.

After signing an informed consent by the patient and, within 24+6 hours following the time of eligibility (time 0), on Day 1, eligible recipient subjects will receive single intravenous (IV) administration of investigational product as described below:

● Allocetra-OTS treatment at 140 x 106 ±20% cells/kg body weight (screening body weight) in 375 mL of Ringer's lactate solution.

Subjects will be followed for efficacy and safety assessments over 28 days following investigational product administration.

Subjects will be hospitalized for COVID-19, and later as medically indicated. Following IP administration (Day 1), subjects will be followed for efficacy and safety assessments through 28 days. The number of visits for subjects participating in this study will be on days 3, 5, 7±1, 14±2, and 28±2. Visits on days 7 and 14 may be done via zoom or telephone.

Study Intervention, Route of Administration, and Dosage Form

Allocetra-OTS is a cell-based therapeutic composed of donor early apoptotic cells.

Patient Classification [National Institutes of Health (NIH)]- www.covid19treatmentguidelines.nih.gov/overview/management-of-covid-19/

In general, adults with COVID-19 can be grouped into the following severity of illness categories:

* Asymptomatic or Pre-symptomatic Infection: Individuals who test positive for SARS-CoV-2 by virologic testing using a molecular diagnostic (e.g., polymerase chain reaction) or antigen test, but have no symptoms.
* Mild Illness: Individuals who have any of the various signs and symptoms of COVID-19 (e.g., fever, cough, sore throat, malaise, headache, muscle pain) without shortness of breath, dyspnea, or abnormal chest imaging.
* Moderate Illness: Individuals who have evidence of lower respiratory disease by clinical assessment or imaging and saturation of oxygen (SpO2) ≥94% on room air at sea level.
* Severe Illness: Individuals who have respiratory frequency >30 breaths per minute, SpO2 <94% on room air at sea level, ratio of arterial partial pressure of oxygen to fraction of inspired oxygen (PaO2/FiO2) <300 mmHg, or lung infiltrates >50%
* Critical Illness: Individuals who have respiratory failure, septic shock, and/or multiple organ dysfunction.

Standard of Care (SOC)

The SOC for COVID-19 will be according to institutional standards. Institutional SOC may include Clexane, anti-viral agents such as Remdesivir, corticosteroids, or other agents.

Concomitant Medications

Prohibited medications: Significant immune-suppressing agents before developing COVID-19, including chronic corticosteroids > 10 mg/day, Azathioprine, Cyclosporine, Cyclophosphamide, and any biological treatment.

The known SOC medications to treat COVID-19; Hydroxychloroquine, Chloroquine, and Azithromycin, are not known to have any possible interaction with Allocetra-OTS. Neither are anti-viral agents.

Concomitant Medical Conditions

Apart from patients with a tumor or end-stage organ condition, chronic diseases like cardiovascular or diabetes are allowed.

ELIGIBILITY:
Inclusion Criteria:

Up to twenty-four subjects, male or female > 18 and < 80-year-old diagnosed with COVID-19, as defined below:

1. Laboratory confirmation of SARS-COV2 infection by reverse-transcription polymerase chain reaction (RT-PCR) from any diagnostic sampling source.
2. Patients classified as severe or critical according to NIH severity classification.
3. All patients will be treated by treating physician with S.C. Clexane, at a minimal dose of 40 mg a day
4. Illness with at least one of the following:

   * Radiographic infiltrates by imaging (chest x-ray, CT scan, etc.), OR
   * SpO2 ≤ 94% on room air, OR
   * Requiring supplemental oxygen, with a P/F ratio of ≤350, ≥150
5. Signed written informed consent by the patient.

Exclusion Criteria:

1. Pregnancy, lactation, and childbearing potential woman who are not willing to use acceptable contraceptives measures for the entire study duration.
2. Combined with other organ failures (need organ support not including respirator), including Stage 4 severe chronic kidney disease or requiring dialysis (i.e. estimated glomerular filtration rate (eGFR) < 30)
3. Patients with a malignant tumor, other serious systemic diseases and psychosis.
4. Patients who are participating in other clinical trials or treated with any experimental agents that may contradict this trial (i.e, biologics)
5. Co-Infection of HIV, tuberculosis.
6. Known immunocompromised state or medications known to be immunosuppressive (see concomitant prohibited medications on the next page).
7. Intubated patients (due to inability to sign an informed consent)
8. Patients with P/F or S/F ratio of <150 or a change in status of eligibility manifested by a rapid decline of P/F ratio between eligibility status and actual drug delivery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Assessment of safety by determining the number of participants with any Adverse Events (AE) and Serious Adverse Events (SAE) | 28 days follow up
  Incidence rates and severity of any Adverse Events (AE) and Serious Adverse Events (SAE)

SECONDARY OUTCOMES:
Preliminary Efficacy: Recovery from COVID-19 as determined by negative PCR or asymptomatic by the NIH classification for the severity of illness | 28 days follow up
  Recovery from COVID-19 will be determined by the following measures:
  The percentage of subjects reporting to 'Asymptomatic' by the NIH classification and the number of days to reach this classification, and/or The percentage of subjects negative for SARS-CoV-2 RNA (by PCR) and the number of days for viral clearance (negative PCR results)
Mortality | 28 days follow up
  Incidence rate of Mortality from any cause
Preliminary Efficacy: To assess prevention of respiratory deterioration associated with COVID-19 by measuring the PaO2/FiO2 ratio | On days, 3, 5, 7, 14, and 28 during 28 days follow up
  Respiratory function will be assessed by measuring the ratio of arterial partial pressure of oxygen to fraction of inspired oxygen (PaO2/FiO2).
  Patients with PaO2/FiO2 ratio < 300mmHg are considered severe patients.
  • The PaO2/FiO2 ratio and its change from the baseline value will be measured on days, 3, 5, 7, 14, and 28.
Hospitalization | 28 days follow up
  Cumulative days in the Intensive care unit (ICU) or COVID-19 ICU or COVID-19 department and/or in hospital.
Life support | 28 days follow up
  Number of ventilator-free days.
Clinical status by the new NIH Patient Classification for the severity of illness | 28 days follow up
  Change from baseline of the new NIH Patient Classification for the severity of illness.
Clinical status by NEWS2 | 28 days follow up
  Change from baseline of National Early Warning Score (NEWS2).
Support measurements: percentage of subjects reporting each severity rating on a 7-point ordinal scale | 28 days follow up
  Percentage of subjects reporting each severity rating on a 7-point ordinal scale at day 28 as follows:
  Death. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO).
  Hospitalized, on non-invasive ventilation or high flow oxygen devices. Hospitalized, requiring supplemental oxygen. Hospitalized, not requiring supplemental oxygen. Not hospitalized, limitation on activities. Not hospitalized, no limitations on activities.
Support measurements: improvement of severity rating on a 7-point ordinal scale | 28 days follow up
  Time to improvement of one category from admission using this 7-point ordinal scale, as follows:
  Death. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO).
  Hospitalized, on non-invasive ventilation or high flow oxygen devices. Hospitalized, requiring supplemental oxygen. Hospitalized, not requiring supplemental oxygen. Not hospitalized, limitation on activities. Not hospitalized, no limitations on activities.
Virus Clearance | Within the 28 days follow up, tested on days 14 and 28
  valuation of clearance of the virus using PCR (Negative for SARS-CoV-2 RNA) on days 14 and 28 (if not negative before).
Exploratory: Serum cytokines/chemokines and immunomodulating factors | 28 days follow up
  Serum concentrations (pg/ml) of cytokines, chemokines, complement, hematopoietic growth factors, and other immunomodulating factors (including HMGB1) will be measured before and after the infusion of Allocetra-OTS and periodically throughout 28 days follow up.
Exploratory: complete blood counts | 28 days follow up
  Differential blood counts will be performed before and after the infusion of Allocetra-OTS and periodically throughout 28 days follow up.
Exploratory: Histone and cell-free DNA levels | 28 days follow up
  Histone and cell-free DNA plasma levels will be measured before and after the infusion of Allocetra-OTS and periodically throughout 28 days follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Dror Mevorach, MD, Principal Investigator — Hadassah Medical Organization; Peter V van Heerden, MD, Principal Investigator — Hadassah Medical Organization
Locations (3):
- Israel (3):
  - Barzilai Medical Center, Ashkelon
  - Hadassah Medical Center, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Heerden PV, Abutbul A, Naama A, Maayan S, Makram N, Nachshon A, Abu Jabal K, Hershkovitz O, Binder L, Shabat Y, Reicher B, Mevorach D. Apoptotic cells for treatment of acute respiratory distress syndrome associated with COVID-19. Front Immunol. 2023 Aug 2;14:1242551. doi: 10.3389/fimmu.2023.1242551. eCollection 2023. PMID 37600829